CLINICAL TRIAL: NCT01980485
Title: The Get Quit-Stay Quit Study: a Randomized Trial of Health Risk Feedback and Relapse Prevention for Treatment-seeking Smokers
Brief Title: The Get Quit - Stay Quit Study
Acronym: GQSQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor of Public Health Sciences and Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37326EP
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Nicotine Dependent Cigarette Smoker
Keywords: smoker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback on lung age and exhaled carbon monoxide (Active Comparator)
  Interventions: Behavioral: Lung Age feedback and exhaled carbon monoxide
- No lung age feedback (Sham Comparator): Those allocated to the control group will simply be informed of their scores on the spirometry.
  Interventions: Behavioral: No Lung Age Feedback

INTERVENTIONS:
Behavioral: Lung Age feedback and exhaled carbon monoxide — In the intervention group, if the lung age is equal to or less than the individual's chronological age, he or she will be briefly informed that the test result was normal and that it is important to avoid potential future lung problems by stopping smoking. For those in the intervention group with a "normal" FEV-1, the intervention will focus on their exhaled carbon-monoxide.
  If their lung age is greater than their chronological age, they will be given their "lung age" in years, and provided with a graph describing the possible decline in lung age if they continued to smoke and a full explanation.
  Those in the Intervention Group will have their exhaled carbon-monoxide (CO) result explained in more detail. Non-smokers typically have an exhaled carbon-monoxide level of 0-4 parts per million, whereas smokers typically have a CO level of 8-50 ppm. CO levels return to normal within a few days of stopping smoking. Participants are provided with a full explanation.
  Arms: Feedback on lung age and exhaled carbon monoxide
Behavioral: No Lung Age Feedback — Those allocated to the control group will simply be informed of their scores on the spirometry.
  Arms: No lung age feedback

SUMMARY:
Narrative: Tobacco smoking remains the single biggest cause of premature death in the United States and the leading cause of cancer and death from cancer. There is therefore an urgent need to find effective but practical ways of helping smokers to quit and stay quit. This randomized trial aims to evaluate two promising methods of helping smokers to quit and to stay quit.

Design: This is a randomized controlled smoking cessation trial with two stages.

In Stage 1, 225 smokers will be recruited and at assessment they will be randomly allocated to receiving feedback on their "Lung Age" as estimated by their Forced Expiratory volume of air from lungs in one second (FEV1), and exhaled carbon-monoxide (CO) (Intervention group 1) or to have these measured but not fed back in a manner designed to enhance motivation to quit (Control group 1). All participants will be provided with group counseling (6 weekly sessions, with the target Quit Date on the day of the second group meeting), and transdermal nicotine patches.

Main outcome measure: Stage 1, Past week tobacco abstinence biochemically validated by exhaled CO < 10 ppm at visit 7 (4 weeks after Target Quit Date).

In Stage 2 (starting visit 7), all participants attending visit 7 (28 days after their Target Quit Date), will be randomly allocated to receiving either the Forever Free relapse prevention materials (Intervention 2) http://www.smokefree.gov/pdf.html or the Surgeon General's Guide "How Tobacco Smoke Causes Disease" (Control 2) http://www.cdc.gov/tobacco/data_statistics/sgr/2010/consumer_booklet/index.htm.

All randomized participants will receive a follow-up phone call a week later to remind them to read and use the materials they have been given, and will attend a follow up visit (8), 6 months after their initial Target Quit Date.

Main outcome measure: Stage 2. Among those who have not smoked in the previous week at visit 7, sustained tobacco abstinence (including no tobacco use in prior 7 days), validated by exhaled CO < 10 ppm at the 6 month visit(8) AND not smoking for any 7 consecutive days during the prior 5 months (definition of a relapse in this study).

Hypothesis: Smokers who are provided with lung age feedback at assessment will have higher quit rates 28 days after the target quit date.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must report smoking at least 5 cigarettes per day for the previous 6 months AND sometimes smoke at least 10 cigarettes in one day.
2. Participants must want to quit smoking and be ready to make a quit attempt within the next 30 days.
3. Participants must plan to remain in the intervention catchment area for at least 8 months.
4. Age >18 years. Nicotine patches are not currently approved by FDA for those under age 18.
5. Participants must be willing to attend and provide data at the 8 study visits, including an assessment visit at which a blood sample will be drawn, 6 group treatment sessions, respond to follow-up telephone calls, and a 6-month follow-up visit.
6. Participants must be able to read and write in English.
7. Nicotine is known to be harmful to the developing human fetus at the recommended therapeutic dose. For this reason women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the standard duration of transdermal nicotine therapy (10 weeks). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating clinician immediately.
8. Ability to understand and the willingness to sign a written informed consent document

   -

Exclusion Criteria:

1. A history of severe allergic reaction while using a nicotine patch.
2. Currently using a drug/medicine as an aid to smoking cessation (e.g. Zyban, Chantix, nicotine replacement).
3. Currently pregnant, trying to get pregnant, or nursing, because nicotine is known to be harmful to the developing human fetus at the recommended therapeutic dose.
4. Had a heart attack, stroke, continuing arrhythmias or angina (chest pains) or abnormal electrocardiogram within the past 4 weeks.
5. Uncontrolled serious mental illness or substance abuse.
6. Uses non-cigarette tobacco products and does not plan to quit all tobacco.

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Penn State Hershey Medical Group Harrisburg, Harrisburg, Pennsylvania
  - Penn State Hershey Medical Group Fishburn Road, Hershey, Pennsylvania
  - Penn State Hershey Internal Medicine, Hershey, Pennsylvania
  - Penn State Hershey Palmyra, Palmyra, Pennsylvania

REFERENCES:
- [Derived] Foulds J, Veldheer S, Hrabovsky S, Yingst J, Sciamanna C, Chen G, Maccani JZ, Berg A. The effect of motivational lung age feedback on short-term quit rates in smokers seeking intensive group treatment: A randomized controlled pilot study. Drug Alcohol Depend. 2015 Aug 1;153:271-7. doi: 10.1016/j.drugalcdep.2015.05.007. Epub 2015 May 18. PMID 26051163

RESULTS

PARTICIPANT FLOW:
Groups:
- Feedback on Lung Age and Exhaled Carbon Monoxide: Lung Age feedback and exhaled carbon monoxide: In the intervention group, if the lung age is equal to or less than the individual's chronological age, he or she will be briefly informed that the test result was normal and that it is important to avoid potential future lung problems by stopping smoking. For those in the intervention group with a "normal" FEV-1, the intervention will focus on their exhaled carbon-monoxide.
  If their lung age is greater than their chronological age, they will be given their "lung age" in years, and provided with a graph describing the possible decline in lung age if they continued to smoke and a full explanation.
  Those in the Intervention Group will have their exhaled carbon-monoxide (CO) result explained in more detail. Non-smokers typically have an exhaled carbon-monoxide level of 0-4 parts per million, whereas smokers typically have a CO level of 8-50 ppm. CO levels return to normal within a few days of stopping smoking. Participants are provided w
Period: Overall Study
Arm/Group | Feedback on Lung Age and Exhaled Carbon Monoxide | No Lung Age Feedback
Started | 120 | 105
Completed | 84 | 80
Not Completed | 36 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Feedback on Lung Age and Exhaled Carbon Monoxide | No Lung Age Feedback | Total
Number analyzed (Participants) | 120 | 105 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 105 | 225
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (12.5) | 49.8 (12.5) | 48.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 72 | 136
  Male | 56 | 33 | 89
Region of Enrollment [Number; unit: participants]
  United States | 120 | 105 | 225

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting no Tobacco Use in the Past 7 Days and Have a Validated CO <10ppm
Description: Exhaled CO <10 ppm and no tobacco use in the past 7 days
Time Frame: 28 days post quit date
Measure: Count of Participants; unit: Participants
Groups:
- Feedback on Lung Age and Exhaled Carbon Monoxide: Lung Age feedback and exhaled carbon monoxide (CO): In the intervention group, if the lung age is equal to or less than the individual's chronological age, he or she will be briefly informed that the test result was normal and that it is important to avoid potential future lung problems by stopping smoking. For those in the intervention group with a "normal" FEV-1, the intervention will focus on their exhaled carbon-monoxide. If their lung age is greater than their chronological age, they will be given their "lung age" in years, and provided with a graph describing the possible decline in lung age if they continued to smoke and a full explanation. Those in the Intervention Group will have their CO result explained in more detail. Non-smokers typically have an exhaled carbon-monoxide level of 0-4 parts per million, whereas smokers typically have a CO level of 8-50 ppm. CO levels return to normal within a few days of stopping smoking. Participants are provided with a full explanation.
Arm/Group | Feedback on Lung Age and Exhaled Carbon Monoxide | No Lung Age Feedback
Number analyzed (Participants) | 120 | 105
Participants | 61 | 55
Statistical Analysis 1: Comparison: Feedback on Lung Age and Exhaled Carbon Monoxide vs No Lung Age Feedback; Test type: Non-Inferiority or Equivalence — This study had 87% power to detect a 40% increase in 28-dayabstinence rates (i.e., from 50% to 70%) based on a two-tailed chi-squared test and alpha = 0.05. We selected this effect size as being at the lower end of the effect size continuum that would be clinically meaningful at 28 days and have the potential to still be meaningful in the longer term even with similar relapse rates in both groups over subsequent months; p = .65, Chi-squared

2. Primary Outcome: Sustained Tobacco Abstinence
Description: Among those who have not smoked in the previous week at visit 7, sustained tobacco abstinence (including no tobacco use in prior 7 days), validated by exhaled CO < 10 ppm at the 6 month visit(8) AND not smoking for any 7 consecutive days during the prior 5 months (definition of a relapse in this study)
Time Frame: 6 months
Population: Those who were quit at 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Forever Free Relapse Materials: Participants received forever free relapse materials
- Surgeon General Brochure: Participants received "A Report from the Surgeon General: How Tobacco Smoke Causes Disease"
Arm/Group | Forever Free Relapse Materials | Surgeon General Brochure
Number analyzed (Participants) | 59 | 56
Participants | 24 | 25

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Feedback on Lung Age and Exhaled Carbon Monoxide | No Lung Age Feedback
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/105
Other Adverse Events (participants affected / at risk) | 25/120 | 24/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Feedback on Lung Age and Exhaled Carbon Monoxide (N=120) | No Lung Age Feedback (N=105)
Flu-like symptoms (General disorders) | 0 | 2
Cardio related (Cardiac disorders) | 3 | 1
Withdrawal Symptoms (Gastrointestinal disorders) | 19 | 13
Respiratory Related (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Other (General disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No